CLINICAL TRIAL: NCT06838247
Title: Detection of Simultaneous Presence of Shoulder Lesions in Patients with Hand Injuries by Diagnostic Ultrasonography
Brief Title: Ultrasonographic Analysis of Post-Traumatic Shoulder Lesions After Hand Trauma
Status: Enrolling by invitation | Type: Observational
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nadide Koca, Principal Investigator, Ankara Training and Research Hospital
Other Study IDs: AnkaraTRH-FTR-NK-02
Record Dates: First submitted 2025-02-16; First posted 2025-02-20 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Shoulder; Ultrasonographic; Hand Injuries
Keywords: Hand injuries; Shoulder; Diagnostic; Ultrasonography
MeSH Terms: conditions — Hand Injuries; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Case: Patients who apply to our hand rehabilitation clinic for rehabilitation after hand injury will undergo routine shoulder examination as well as hand examination. The group with shoulder symptoms and examination findings will constitute the case group.
- Control: The group with a normal shoulder examination and ultrasonographic findings will be the control group.

SUMMARY:
The purpose of the study is to reveal whether there are concurrent shoulder lesions in patients with hand injuries. Its importance is that it will shed light on whether not only the hand but also the shoulder should be included in the treatment program in hand rehabilitation.

DETAILED DESCRIPTION:
Hand injuries constitute one fifth of the injuries that are brought to the emergency room and one third of the work accidents. They are very costly because they require surgical intervention and a long rehabilitation process and delay the patient's return to work. The general tendency in hand rehabilitation is to focus more on treatments focused on the hand and wrist.

There are studies that draw attention to the relationship between hand grip strength and rotator cuff function and that other upper extremity musculoskeletal injuries are often neglected in patients with hand injuries. This may affect rehabilitation results and prevent the patient from returning to daily activities.

It is reported that in patients with hand and wrist injuries, other upper extremity musculoskeletal problems are seen simultaneously in 40% of cases and most of these are related to the shoulder.

It is reported that rotator cuff problems and lateral epicondylitis are 9 times more common even in carpal tunnel syndrome, which is a relatively simple hand problem that is encountered very frequently in clinical practice.

Traumatic hand injuries can also affect all upper extremity functions. In these patients, it was determined that there was weakness in both the ipsilateral supraspinatus and infraspinatus muscles. The researchers emphasized that the inclusion of shoulder muscle training during the postoperative rehabilitation protocol and selective strengthening of the rotator cuff muscles in distal extremity problems may be clinically important.

In studies conducted to detect shoulder problems in patients with hand injuries, either patient examination or self-reports of the patients have been used so far.

In this study, the investigators aimed to concretely reveal shoulder pathologies by evaluating the results of diagnostic ultrasonography performed on our patients with shoulder symptoms. In this way, the investigators aimed to obtain a clearer result on whether the shoulder should be included in the hand rehabilitation program.

Our study is the first study to evaluate shoulder pathologies in patients with hand injuries with diagnostic ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* Having a history of hand injury and applying for hand rehabilitation after surgical and conservative treatment.

Exclusion Criteria:

* Being under 18 and over 65 years of age
* Patients with systemic diseases (Diabetes mellitus, Peripheral vascular diseases)
* Any rheumatic disease involving the hand and upper extremity
* History of neuropathy involving the hand and upper extremity
* Those with any shoulder problems prior to the hand injury
* Those with an open wound on the hand
* Those who cannot cooperate
* Other upper extremity traumatic injuries occurring during the hand injury

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who apply to our hand rehabilitation clinic for rehabilitation after hand injury will undergo a routine shoulder examination as well as a hand examination. The group with shoulder symptoms and examination findings will constitute the case group, and the group with a normal shoulder examination will constitute the control group. Age, gender, height, weight, occupation, dominant hand, type of injury, type of injury, duration of injury, operation time, and immobilization time will be recorded for both groups.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-04-16 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic shoulder ultrasonography | up to 12 weeks
  For shoulder ultrasonography, the specialist physician and the patient will sit opposite each other. The examination will be performed using high-resolution linear probes. Standard ultrasonography technique and diagnosis will be used, and real-time ultrasonography will be performed with an ultrasound device with a 6-11 MHz linear wide-band probe (Nemio XH, Toshiba, Japan). In shoulder ultrasonography, the long head of the biceps brachialis muscle, supraspinatus tendon and subacromial bursa will be examined. Fluid increase or edema in the subacromial bursa will be evaluated to determine whether there is subacromial bursitis. In case of suspected supraspinatus tendon rupture, the contour integrity, echogenicity and thickness of the tendon will be carefully examined; in addition, it will be determined whether there is a partial or complete tear on the tendon.

SECONDARY OUTCOMES:
Visual analog scale (VAS) scores | up to 12 weeks
  VAS is used to convert some values that cannot be measured quantitatively into numerical values. In VAS, where pain intensity is evaluated, pain intensity is graded between 0 and 10 points. "No pain" is graded as 0 points and "very severe pain" is graded as 10 points. Pain intensity of "less than 3 points" is indicated as mild pain, "between 3-6 points" as moderate pain, and "more than 6 points" as severe pain.
  Visual pain scoring will be done separately for both the hand and shoulder regions.
Joint range of motion | up to 12 weeks
  Joint range of motion is known as ROM and refers to the measurement of the amount of movement around a specific joint. Joint range of motion will be measured with the help of a tool called a goniometer. Joint range of motion will be measured and recorded in both the hand joint and shoulder joint.
Handgrip Strength Test | up to 12 weeks
  Grip strength is a measure of muscle strength or the maximum force/tension produced by a person's forearm muscles. It can be used as a screening tool for measuring upper body strength and general strength. Grip strength will be assessed with a Jamar dynamometer and the values obtained will be recorded.
The Shoulder Pain and Disability Index | up to 12 weeks
  The Shoulder Pain and Disability Index (SPADI) is a 13-item questionnaire divided into pain and activity limitation categories. It focuses on the degree of pain or disability caused by shoulder problems in the past week. The patient answers the questions himself/herself using a VAS or NRS scale. The higher a patient scores on the SPADI, the greater the pain/limitation in activities.
  The score for each subscale is obtained by adding all individual scores for the subscale and dividing the result by the maximum score for the subscale. The normalized score is converted to a scale of 0 to 100, with 100 indicating severe problems and 0 indicating no problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy and Rehabilitation, University of Health Sciences, Ankara Training and Research Hospital, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdallah EA, Eldesoky MT, Saweres JW, Abdelhaleem MD. Effect of Adding Shoulder Stabilization Exercises to the Rehabilitation of Postoperative Hand Injuries in Young Adult Patients. Hand (N Y). 2025 Jul;20(5):778-784. doi: 10.1177/15589447241232017. Epub 2024 Feb 15. PMID 38357889
- [Background] Winiarski LM, Livoni JD, Madsen PV, Rathleff MS, Larsen P. Concurrent musculoskeletal complaints in elbows, shoulders, and necks after common hand and forearm injuries or conditions: A cross-sectional study among 600 patients. J Hand Ther. 2021 Oct-Dec;34(4):543-548. doi: 10.1016/j.jht.2020.05.002. Epub 2020 Sep 4. PMID 32893097
- [Background] Horsley I, Herrington L, Hoyle R, Prescott E, Bellamy N. Do changes in hand grip strength correlate with shoulder rotator cuff function? Shoulder Elbow. 2016 Apr;8(2):124-9. doi: 10.1177/1758573215626103. Epub 2016 Jan 25. PMID 27583010
- [Background] Xue R, Wong J, Imere A, King H, Clegg P, Cartmell S. Current clinical opinion on surgical approaches and rehabilitation of hand flexor tendon injury-a questionnaire study. Front Med Technol. 2024 Feb 15;6:1269861. doi: 10.3389/fmedt.2024.1269861. eCollection 2024. PMID 38425421
- [Background] Jha CK, Shukla Y, Mukherjee R, Rathva P, Joshi M, Jain D. A Glove-Based Virtual Hand Rehabilitation System for Patients With Post-Traumatic Hand Injuries. IEEE Trans Biomed Eng. 2024 Jul;71(7):2033-2041. doi: 10.1109/TBME.2024.3360888. Epub 2024 Jun 19. PMID 38294922